CLINICAL TRIAL: NCT03519737
Title: A Phase 3, Randomized, Placebo-Controlled, Double-Blind Study of the Aureva Transcranial Ultrasound Device With Tissue Plasminogen Activator in Patients With Acute Ischemic Stroke (TRUST)
Brief Title: Aureva Transcranial Ultrasound Device With tPA in Patients With Acute Ischemic Stroke
Acronym: TRUST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cerevast Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM-CP-01
Record Dates: First submitted 2018-04-17; First posted 2018-05-09 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke; Acute Stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Intervention Model Description: Sham control and active insonation. During lead-in phase for the first 40 subjects, only active insonation will be programmed.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding is achieved through operator entry of a randomization variable obtained from IWRS at the time of enrollment and randomization. This randomization variable (A or B), the meaning of which is blinded to the operator, is entered into the control box and determines the mode of the device as either active insonation or sham insonation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Control group (tPA + sham TUS) (Sham Comparator): Control group (tPA + sham TUS) During the primary phase of the study, subjects will be randomized 1:1
  Interventions: Device: tPA in combination with the Sonolysis Headframe (Sham TUS)
- Treatment group (tPA + TUS) (Active Comparator): Treatment group (tPA + TUS): Lead-in phase and Primary phase
  Interventions: Device: tPA in combination with the Sonolysis Headframe (TUS)

INTERVENTIONS:
Device: tPA in combination with the Sonolysis Headframe (TUS) — tPA: 60 minutes per approved labeling TUS insonation via the Sonolysis Headframe: minimum 90 minutes - maximum 120 minutes
  Other Names: Aureva Headframe (TUS) with Tissue Plaminogen Activator (tPA)
  Arms: Treatment group (tPA + TUS)
Device: tPA in combination with the Sonolysis Headframe (Sham TUS) — tPA per approved labeling Sham (inactive) TUS insonation via the Sonolysis Headframe: minimum 90 minutes - maximum 120 minutes
  Other Names: Aureva Headframe (Sham TUS) with Tissue Plaminogen Activator (tPA)
  Arms: Control group (tPA + sham TUS)

SUMMARY:
This is a randomized, placebo controlled, double-blind phase 3 clinical study to evaluate the efficacy and safety of transcranial ultrasound (TUS) using the Sonolysis Headframe as an adjunctive therapy to intravenous (IV) tissue plasminogen activator (tPA) therapy in subjects with acute ischemic stroke that initially present at non-endovascular (EVT) treating hospitals that have established transport services in place to transfer subjects to hospitals capable of performing EVT.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the safety and efficacy of TUS using the Sonolysis Headframe in combination with systemic tPA (Treatment group) compared to systemic tPA alone (Control group) in subjects with acute ischemic stroke.

Number of Subjects Required:

Lead-in Phase: 40 subjects in the U.S.; Primary Phase: 556 total enrolled subjects (278 per arm)

Number of Study Centers:

Lead-in Phase: Up to 20 Institutions in U.S.; Primary Phase: Up to 70 Institutions worldwide

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with acute ischemic stroke
2. Subjects that initially present at non-EVT treating hospitals that have established transport services in place to transfer subjects to hospitals capable of performing EVT
3. Males or females 18 - 80 years of age
4. Subjects presenting within time window for IV tPA treatment approved by local regulatory authorities but no more than 4.5 hours from onset of symptoms
5. No signs of intracranial bleeding on assessment by non-contrast CT
6. Subjects that in the opinion of the treating physician require treatment with full dose of IV tPA (0.9mg/kg) as standard of care per institutional standards
7. SBP ≤ 185 mmHg and DBP ≤ 105 mmHg at baseline or after treatment of hypertension with medications prior to tPA bolus
8. Pre-morbid mRS of 0-1
9. Arterial occlusion in the middle cerebral artery (MCA) M1 or proximal M2, intracranial carotid T, anterior cerebral artery (ACA) A1, basilar, proximal posterior cerebral artery (PCA) P1 or intracranial tandem lesions in these locations visible on CT angiography (CTA)
10. Provision of informed consent as demonstrated by the subject's signature or by the signature of the subject's authorized legal representative on the Informed Consent Form in accordance with all local and national regulations and no later than 15 minutes after standard of care tPA administration

Exclusion Criteria:

1. Tandem lesions where one lesion is extracranial (carotid or vertebral artery)
2. ASPECTS score < 6 on non contrast CT or ischemic changes that in the opinion of the investigator would be medically inappropriate for reperfusion therapy
3. Poor collateral circulation defined as minimal or no pial collaterals in >50% of the ischemic territory
4. Expected time between activation of Sonolysis Headframe and initiation of EVT < 90 minutes
5. Pregnant or breast feeding women, clinical signs of pericarditis, sepsis or any other serious medical illness likely to interact with treatment, confounding preexistent neurological or psychiatric disease or test values that, in the opinion of the investigator, pose significant risk to the subject and warrant exclusion from the study
6. Impaired renal function defined as eGFR < 60 mL/min/1.73 m2
7. No permanent address or phone number
8. Any investigational drug <14 days prior to study participation
9. Subjects with known allergy to x-ray contrast material
10. Subjects with any standard contraindication for intravenous tPA therapy as per local or national guidelines

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Estimated)
Dates: Start 2018-08-17 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete recanalization measured by modified Arterial Occlusive Lesion (mAOL) | 90-120 minutes post TUS treatment before EVT
  Complete recanalization of the primary occluded vessel as measured by the modified Arterial Occlusive Lesion (mAOL) scoring system. The mAOL assigns a score from 0 to 3, which represents the range from no recanalization to complete recanalization based on either the presence (grade 2 or 3) or absence (grades 0 or 1) of any downstream flow.

SECONDARY OUTCOMES:
modified Rankin Scale (mRS) score 0-2 | 90 days +/- 10 days
  Functional dependence at 90 days as measured by the modified Rankin Scale (mRS). The mRS consists of 7 grades, (0-6), with 0 corresponding to no symptoms and 6 corresponding to death. For this study, functional independence will be defined as those subjects that achieve a mRS score of 0-2 at 90 days.
Neurologic Status at 24 hours post treatment measured by National Institute of Health's Stroke Scale (NIHSS). | 24 hours post TUS treatment
  NIHSS has 15 items. Ratings for each item are scored on a 0-3 to 0-5 scale, with a total score of 0 for normal and 42 for maximally impaired.
Partial or complete recanalization as measured by mAOL score of 2-3. | 90-120 minutes post TUS treatment before EVT
  See description in Primary Outcome Measure.
Partial or complete recanalization as measured by Thrombolysis In Cerebral Ischemia (TICI) score of 2-3 | 90-120 minutes post TUS treatment before EVT
  TICI Scale: [0] - No antegrade flow beyond the point of occlusion. [1] - The contrast material passes beyond the area of obstruction but fails to opacify the entire cerebral bed distal to the obstruction. [2] - The contrast material passes beyond the obstruction and opacifies the arterial bed distal to the obstruction. However, the rate of entry of contrast into the vessel distal to the obstruction and/or its rate of clearance from the distal bed are perceptibly slower than its entry into and/or clearance from comparable areas not perfused by the previously occluded vessel. [3] - Antegrade flow into the bed distal to the obstruction occurs as promptly as into the obstruction and clearance of contrast material from the involved bed is as rapid as from an uninvolved other bed of the same vessel or the opposite cerebral artery.

CONTACTS AND LOCATIONS:
Overall Officials: Andrei V Alexandrov, MD, Principal Investigator — University of Tennessee
Locations (2):
- United States (2):
  - The University of Tennessee Health Science Center, Memphis, Tennessee
  - Memorial Hermann Hospital - Texas Medical Center (TMC), Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Writing Group Members; Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, Das SR, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Isasi CR, Jimenez MC, Judd SE, Kissela BM, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Magid DJ, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Rosamond W, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee; Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2016 Update: A Report From the American Heart Association. Circulation. 2016 Jan 26;133(4):e38-360. doi: 10.1161/CIR.0000000000000350. Epub 2015 Dec 16. No abstract available. PMID 26673558
- [Background] National Institute of Neurological Disorders and Stroke rt-PA Stroke Study Group. Tissue plasminogen activator for acute ischemic stroke. N Engl J Med. 1995 Dec 14;333(24):1581-7. doi: 10.1056/NEJM199512143332401. PMID 7477192
- [Background] Zivin JA. Acute stroke therapy with tissue plasminogen activator (tPA) since it was approved by the U.S. Food and Drug Administration (FDA). Ann Neurol. 2009 Jul;66(1):6-10. doi: 10.1002/ana.21750. PMID 19681102
- [Background] Gravanis I, Tsirka SE. Tissue-type plasminogen activator as a therapeutic target in stroke. Expert Opin Ther Targets. 2008 Feb;12(2):159-70. doi: 10.1517/14728222.12.2.159. PMID 18208365
- [Background] Mishra SM, Dykeman J, Sajobi TT, Trivedi A, Almekhlafi M, Sohn SI, Bal S, Qazi E, Calleja A, Eesa M, Goyal M, Demchuk AM, Menon BK. Early reperfusion rates with IV tPA are determined by CTA clot characteristics. AJNR Am J Neuroradiol. 2014 Dec;35(12):2265-72. doi: 10.3174/ajnr.A4048. Epub 2014 Jul 24. PMID 25059699
- [Background] Bhatia R, Hill MD, Shobha N, Menon B, Bal S, Kochar P, Watson T, Goyal M, Demchuk AM. Low rates of acute recanalization with intravenous recombinant tissue plasminogen activator in ischemic stroke: real-world experience and a call for action. Stroke. 2010 Oct;41(10):2254-8. doi: 10.1161/STROKEAHA.110.592535. Epub 2010 Sep 9. PMID 20829513
- [Background] Raychev R, Saver JL. Mechanical thrombectomy devices for treatment of stroke. Neurol Clin Pract. 2012 Sep;2(3):231-235. doi: 10.1212/CPJ.0b013e31826af206. PMID 23634369
- [Background] Broderick JP, Palesch YY, Demchuk AM, Yeatts SD, Khatri P, Hill MD, Jauch EC, Jovin TG, Yan B, Silver FL, von Kummer R, Molina CA, Demaerschalk BM, Budzik R, Clark WM, Zaidat OO, Malisch TW, Goyal M, Schonewille WJ, Mazighi M, Engelter ST, Anderson C, Spilker J, Carrozzella J, Ryckborst KJ, Janis LS, Martin RH, Foster LD, Tomsick TA; Interventional Management of Stroke (IMS) III Investigators. Endovascular therapy after intravenous t-PA versus t-PA alone for stroke. N Engl J Med. 2013 Mar 7;368(10):893-903. doi: 10.1056/NEJMoa1214300. Epub 2013 Feb 7. PMID 23390923
- [Background] Kidwell CS, Jahan R, Gornbein J, Alger JR, Nenov V, Ajani Z, Feng L, Meyer BC, Olson S, Schwamm LH, Yoo AJ, Marshall RS, Meyers PM, Yavagal DR, Wintermark M, Guzy J, Starkman S, Saver JL; MR RESCUE Investigators. A trial of imaging selection and endovascular treatment for ischemic stroke. N Engl J Med. 2013 Mar 7;368(10):914-23. doi: 10.1056/NEJMoa1212793. Epub 2013 Feb 8. PMID 23394476
- [Background] Ciccone A, Valvassori L, Nichelatti M, Sgoifo A, Ponzio M, Sterzi R, Boccardi E; SYNTHESIS Expansion Investigators. Endovascular treatment for acute ischemic stroke. N Engl J Med. 2013 Mar 7;368(10):904-13. doi: 10.1056/NEJMoa1213701. Epub 2013 Feb 6. PMID 23387822
- [Background] Berkhemer OA, Fransen PS, Beumer D, van den Berg LA, Lingsma HF, Yoo AJ, Schonewille WJ, Vos JA, Nederkoorn PJ, Wermer MJ, van Walderveen MA, Staals J, Hofmeijer J, van Oostayen JA, Lycklama a Nijeholt GJ, Boiten J, Brouwer PA, Emmer BJ, de Bruijn SF, van Dijk LC, Kappelle LJ, Lo RH, van Dijk EJ, de Vries J, de Kort PL, van Rooij WJ, van den Berg JS, van Hasselt BA, Aerden LA, Dallinga RJ, Visser MC, Bot JC, Vroomen PC, Eshghi O, Schreuder TH, Heijboer RJ, Keizer K, Tielbeek AV, den Hertog HM, Gerrits DG, van den Berg-Vos RM, Karas GB, Steyerberg EW, Flach HZ, Marquering HA, Sprengers ME, Jenniskens SF, Beenen LF, van den Berg R, Koudstaal PJ, van Zwam WH, Roos YB, van der Lugt A, van Oostenbrugge RJ, Majoie CB, Dippel DW; MR CLEAN Investigators. A randomized trial of intraarterial treatment for acute ischemic stroke. N Engl J Med. 2015 Jan 1;372(1):11-20. doi: 10.1056/NEJMoa1411587. Epub 2014 Dec 17. PMID 25517348
- [Background] Goyal M, Demchuk AM, Menon BK, Eesa M, Rempel JL, Thornton J, Roy D, Jovin TG, Willinsky RA, Sapkota BL, Dowlatshahi D, Frei DF, Kamal NR, Montanera WJ, Poppe AY, Ryckborst KJ, Silver FL, Shuaib A, Tampieri D, Williams D, Bang OY, Baxter BW, Burns PA, Choe H, Heo JH, Holmstedt CA, Jankowitz B, Kelly M, Linares G, Mandzia JL, Shankar J, Sohn SI, Swartz RH, Barber PA, Coutts SB, Smith EE, Morrish WF, Weill A, Subramaniam S, Mitha AP, Wong JH, Lowerison MW, Sajobi TT, Hill MD; ESCAPE Trial Investigators. Randomized assessment of rapid endovascular treatment of ischemic stroke. N Engl J Med. 2015 Mar 12;372(11):1019-30. doi: 10.1056/NEJMoa1414905. Epub 2015 Feb 11. PMID 25671798
- [Background] Campbell BC, Mitchell PJ, Kleinig TJ, Dewey HM, Churilov L, Yassi N, Yan B, Dowling RJ, Parsons MW, Oxley TJ, Wu TY, Brooks M, Simpson MA, Miteff F, Levi CR, Krause M, Harrington TJ, Faulder KC, Steinfort BS, Priglinger M, Ang T, Scroop R, Barber PA, McGuinness B, Wijeratne T, Phan TG, Chong W, Chandra RV, Bladin CF, Badve M, Rice H, de Villiers L, Ma H, Desmond PM, Donnan GA, Davis SM; EXTEND-IA Investigators. Endovascular therapy for ischemic stroke with perfusion-imaging selection. N Engl J Med. 2015 Mar 12;372(11):1009-18. doi: 10.1056/NEJMoa1414792. Epub 2015 Feb 11. PMID 25671797
- [Background] Saver JL, Goyal M, Bonafe A, Diener HC, Levy EI, Pereira VM, Albers GW, Cognard C, Cohen DJ, Hacke W, Jansen O, Jovin TG, Mattle HP, Nogueira RG, Siddiqui AH, Yavagal DR, Baxter BW, Devlin TG, Lopes DK, Reddy VK, du Mesnil de Rochemont R, Singer OC, Jahan R; SWIFT PRIME Investigators. Stent-retriever thrombectomy after intravenous t-PA vs. t-PA alone in stroke. N Engl J Med. 2015 Jun 11;372(24):2285-95. doi: 10.1056/NEJMoa1415061. Epub 2015 Apr 17. PMID 25882376
- [Background] Jovin TG, Chamorro A, Cobo E, de Miquel MA, Molina CA, Rovira A, San Roman L, Serena J, Abilleira S, Ribo M, Millan M, Urra X, Cardona P, Lopez-Cancio E, Tomasello A, Castano C, Blasco J, Aja L, Dorado L, Quesada H, Rubiera M, Hernandez-Perez M, Goyal M, Demchuk AM, von Kummer R, Gallofre M, Davalos A; REVASCAT Trial Investigators. Thrombectomy within 8 hours after symptom onset in ischemic stroke. N Engl J Med. 2015 Jun 11;372(24):2296-306. doi: 10.1056/NEJMoa1503780. Epub 2015 Apr 17. PMID 25882510
- [Background] Alexandrov AV, Molina CA, Grotta JC, Garami Z, Ford SR, Alvarez-Sabin J, Montaner J, Saqqur M, Demchuk AM, Moye LA, Hill MD, Wojner AW; CLOTBUST Investigators. Ultrasound-enhanced systemic thrombolysis for acute ischemic stroke. N Engl J Med. 2004 Nov 18;351(21):2170-8. doi: 10.1056/NEJMoa041175. PMID 15548777
- [Background] Tsivgoulis G, Eggers J, Ribo M, Perren F, Saqqur M, Rubiera M, Sergentanis TN, Vadikolias K, Larrue V, Molina CA, Alexandrov AV. Safety and efficacy of ultrasound-enhanced thrombolysis: a comprehensive review and meta-analysis of randomized and nonrandomized studies. Stroke. 2010 Feb;41(2):280-7. doi: 10.1161/STROKEAHA.109.563304. Epub 2009 Dec 31. PMID 20044531
- [Background] Sakharov DV, Rijken DC. The effect of flow on lysis of plasma clots in a plasma environment. Thromb Haemost. 2000 Mar;83(3):469-74. PMID 10744155
- [Background] Guo T, Li H, Lv Y, Lu H, Niu J, Sun J, Yang GY, Ren C, Tong S. Pulsed Transcranial Ultrasound Stimulation Immediately After The Ischemic Brain Injury is Neuroprotective. IEEE Trans Biomed Eng. 2015 Oct;62(10):2352-7. doi: 10.1109/TBME.2015.2427339. Epub 2015 Apr 28. PMID 25935023
- [Background] Alexandrov AV, Barlinn K, Strong R, Alexandrov AW, Aronowski J. Low-Power 2-MHz Pulsed-Wave Transcranial Ultrasound Reduces Ischemic Brain Damage in Rats. Transl Stroke Res. 2011 Sep;2(3):376-81. doi: 10.1007/s12975-011-0080-6. Epub 2011 Apr 21. PMID 24323655
- [Background] Barreto AD, Alexandrov AV, Shen L, Sisson A, Bursaw AW, Sahota P, Peng H, Ardjomand-Hessabi M, Pandurengan R, Rahbar MH, Barlinn K, Indupuru H, Gonzales NR, Savitz SI, Grotta JC. CLOTBUST-Hands Free: pilot safety study of a novel operator-independent ultrasound device in patients with acute ischemic stroke. Stroke. 2013 Dec;44(12):3376-81. doi: 10.1161/STROKEAHA.113.002713. Epub 2013 Oct 24. PMID 24159060
- [Background] Khatri P, Neff J, Broderick JP, Khoury JC, Carrozzella J, Tomsick T; IMS-I Investigators. Revascularization end points in stroke interventional trials: recanalization versus reperfusion in IMS-I. Stroke. 2005 Nov;36(11):2400-3. doi: 10.1161/01.STR.0000185698.45720.58. Epub 2005 Oct 13. PMID 16224088
- [Background] Zaidat OO, Yoo AJ, Khatri P, Tomsick TA, von Kummer R, Saver JL, Marks MP, Prabhakaran S, Kallmes DF, Fitzsimmons BF, Mocco J, Wardlaw JM, Barnwell SL, Jovin TG, Linfante I, Siddiqui AH, Alexander MJ, Hirsch JA, Wintermark M, Albers G, Woo HH, Heck DV, Lev M, Aviv R, Hacke W, Warach S, Broderick J, Derdeyn CP, Furlan A, Nogueira RG, Yavagal DR, Goyal M, Demchuk AM, Bendszus M, Liebeskind DS; Cerebral Angiographic Revascularization Grading (CARG) Collaborators; STIR Revascularization working group; STIR Thrombolysis in Cerebral Infarction (TICI) Task Force. Recommendations on angiographic revascularization grading standards for acute ischemic stroke: a consensus statement. Stroke. 2013 Sep;44(9):2650-63. doi: 10.1161/STROKEAHA.113.001972. Epub 2013 Aug 6. No abstract available. PMID 23920012
- [Background] Jung C, Yoon W, Ahn SJ, Choi BS, Kim JH, Suh SH. The Revascularization Scales Dilemma: Is It Right to Apply the Treatment in Cerebral Ischemia Scale in Posterior Circulation Stroke? AJNR Am J Neuroradiol. 2016 Feb;37(2):285-9. doi: 10.3174/ajnr.A4529. Epub 2015 Sep 17. PMID 26381554
- [Background] Higashida RT, Furlan AJ, Roberts H, Tomsick T, Connors B, Barr J, Dillon W, Warach S, Broderick J, Tilley B, Sacks D; Technology Assessment Committee of the American Society of Interventional and Therapeutic Neuroradiology; Technology Assessment Committee of the Society of Interventional Radiology. Trial design and reporting standards for intra-arterial cerebral thrombolysis for acute ischemic stroke. Stroke. 2003 Aug;34(8):e109-37. doi: 10.1161/01.STR.0000082721.62796.09. Epub 2003 Jul 17. PMID 12869717